CLINICAL TRIAL: NCT06969521
Title: Online Assessment and Enhancement of Auditory Perception for Speech Sound Errors: Online Rotating Delivery of Perception/Production Enhanced Treatment for Rhotics
Brief Title: Online Rotating Delivery of Perception/Production Enhanced Treatment for Rhotics
Acronym: ORDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montclair State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20-21-2137-Study 4; 2R15DC019775-02 (NIH)
Record Dates: First submitted 2025-04-22; First posted 2025-05-14 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Speech Sound Disorder
Keywords: speech sound disorder; auditory perception; articulation
MeSH Terms: conditions — Speech Sound Disorder

STUDY DESIGN:
Intervention Model Description: Children with RSSD may vary in pre-treatment speech production severity, and the extent to which they can approximate /r/ may be an important indicator of subsequent treatment response. In addition, perceptual acuity may influence how participants respond to perception and/or production treatment. Therefore, a blocked randomization procedure will be used to protect against a situation where treatment groups are unbalanced with respect to pre-treatment severity in either the perception or production domain. Based on the treating clinicians' perceptual ratings of participants' performance in /r/ word probes administered in the pre-treatment evaluation phase, participants will be categorized as High Accuracy (>10% accuracy) or Low Accuracy (<=10% accuracy), a cutoff determined from pre-treatment baseline data aggregated over 11 studies previously conducted by our team. We will henceforth refer to these groups as "production accuracy groups." In addition, we will use the criteria adopted i
Who Masked: Outcomes Assessor
Masking Description: All perceptual ratings will be obtained from blinded, skilled clinician listeners recruited and trained in previous studies. Following protocols refined in previous published research, binary rating responses (1=correct; 0=incorrect) will be aggregated over at least 4 unique listeners per token.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ORDER: Visual acoustic biofeedback training (Active Comparator): The investigators will use the following approach, adopted successfully for the RCT in the previous funding cycle:
  (1) Participants will be randomized after providing informed consent, meeting eligibility requirements, and completing the tasks and clinician-rated baselines that determine response group (High, Low). (2) For each perception accuracy group, the statistician will develop 2 batches of 10 concealed envelopes for assignment, one for high production accuracy participants and one for low production accuracy participants. Each will contain 10 participant assignments in random order: 5 TAU+ Perception-first, 5 TAU-first. Thus, once the investigators have recruited the first 10 participants for one subgroup (e.g., Low Perceptual Accuracy, Low Production Accuracy), another batch of 10 envelopes will be generated to allocate the next 10 children recruited in that subgroup.
  Interventions: Behavioral: Visual acoustic biofeedback: ORDER
- ORDER: Perceptual training (Experimental): The investigators will use the following approach, adopted successfully for the RCT in the previous funding cycle: (1) Participants will be randomized after providing informed consent, meeting eligibility requirements, and completing the tasks and clinician-rated baselines that determine response group (High, Low). (2) For each perception accuracy group, the statistician will develop 2 batches of 10 concealed envelopes for assignment, one for high production accuracy participants and one for low production accuracy participants. Each will contain 10 participant assignments in random order: 5 TAU+ Perception-first, 5 TAU-first. Thus, once we have recruited the first 10 participants for one subgroup (e.g., Low Perceptual Accuracy, Low Production Accuracy), another batch of 10 envelopes will be generated to allocate the next 10 children recruited in that subgroup.
  Interventions: Behavioral: Perception Training: ORDER
- ORDER: No treatment (No Intervention): No treatment, 4-week period of no treatment

INTERVENTIONS:
Behavioral: Visual acoustic biofeedback: ORDER — In visual-acoustic biofeedback treatment, elements of traditional articulation treatment are used, including auditory models, verbal descriptions of correct articulator placement, cues for repetitive motor practice via images and diagrams of the vocal tract as visual aids. These strategies are supplemented with a dynamic display of the speech signal in the form of the real-time LPC (Linear Predictive Coding) spectrum (Sona-Match module of PENTAX Sona- Speech software). Because correct vs incorrect productions of /r/ contrast acoustically in the frequency of the third formant (F3), participants will be cued to make their real-time LPC spectrum match a visual target characterized by a low F3 frequency. They will be encouraged to attend to the visual display while adjusting the placement of their articulators and observing how those adjustments impact F3. Knowledge of performance feedback will typically involve reference to the location of the third peak on the visual display.
  Arms: ORDER: Visual acoustic biofeedback training
Behavioral: Perception Training: ORDER — Description: Perceptual training involves self-paced presentation of auditory stimuli via a computerized software program (Gorilla). Stimuli are organized into three separate tasks. In tasks 1 and 3, which train category goodness judgment, participants will hear 75 naturally produced speech tokens containing /r/ from various speakers, with a balance of correct and incorrect productions. They will classify each /r/ as correct or incorrect and receive feedback on the accuracy of their classification. Tasks 1 and 3 differ in that task 1 will feature a subset of items designed to provide focused practice on a specific context (e.g., initial /r/ as in red; /r/ as syllable nucleus as in sir), with increasing difficulty over time, whereas task 3 will feature randomly selected items representing all contexts and difficulty levels. In task 2, participants will hear 75 items drawn from the synthetic rake-wake continuum used in the identification task administered at baseline, but they will recei
  Arms: ORDER: Perceptual training

SUMMARY:
The goal of this clinical trial is to determine whether perceptual training enhances speech perception and production outcomes in children with Residual Speech Sound Disorders (RSSD). The main questions it aims to answer are:

Does pre-treatment speech production accuracy predict treatment response?

Does perceptual acuity influence the effectiveness of perception-first versus production-first interventions?

Researchers will compare TAU+Perception-first and TAU-first treatment conditions to see if the order of intervention affects speech improvement outcomes, particularly based on participants' initial perception and production accuracy.

Participants will:

Complete pre-treatment evaluations to assess /r/ production and speech perception.

Be grouped into high or low production and perception accuracy categories based on established thresholds.

Be randomly assigned (using a blocked randomization procedure) to one of two treatment arms via telepractice.

Participate in the assigned treatment condition designed to target speech sound accuracy.

Randomization is stratified to ensure treatment groups are balanced based on pre-treatment severity in both the perception and production domains.

DETAILED DESCRIPTION:
Children with RSSD may vary in pre-treatment speech production severity, and the extent to which they can approximate /r/ may be an important indicator of subsequent treatment response. In addition, perceptual acuity may influence how participants respond to perception and/or production treatment. Therefore, a blocked randomization procedure will be used to protect against a situation where treatment groups are unbalanced with respect to pre-treatment severity in either the perception or production domain. Based on the treating clinicians' perceptual ratings of participants' performance in /r/ word probes administered in the pre-treatment evaluation phase, participants will be categorized as High Accuracy (>10% accuracy) or Low Accuracy (<=10% accuracy), a cutoff determined from pre-treatment baseline data aggregated over 11 studies previously conducted by our team. The investigators will henceforth refer to these groups as "production accuracy groups." In addition, the investigators will use the criteria adopted in the previous funding cycle to classify participants into high or low perception groups (henceforth, "perception accuracy groups"). Participants will be randomized to the TAU(Treatment as Usual) +Perception-first or TAU-first condition via telepractice with stratification on both perception and production accuracy group. Randomization will be supervised by statistician J. Hill at the NYU site. The investigators will use the following approach, adopted successfully for the RCT in the previous funding cycle: (1) Participants will be randomized after providing informed consent, meeting eligibility requirements, and completing the tasks and clinician-rated baselines that determine response group (High, Low). (2) For each perception accuracy group, the statistician will develop 2 batches of 10 concealed envelopes for assignment, one for high production accuracy participants and one for low production accuracy participants. Each will contain 10 participant assignments in random order: 5 TAU+ Perception-first, 5 TAU-first. (3) The investigators cannot fully predict the exact proportion of participants with high versus low production accuracy in each category of perceptual accuracy, so it is possible that the investigators will encounter significantly more in one group than the other. Thus, once the investigators have recruited the first 10 participants for one subgroup (e.g., Low Perceptual Accuracy, Low Production Accuracy), another batch of 10 envelopes will be generated to allocate the next 10 children recruited in that subgroup.

ELIGIBILITY:
Inclusion Criteria:

Must be between 8;0 and 17;11 years of age at the time of enrollment. Must speak English as the dominant language (i.e., must have begun learning English by age 2, per parent report).

Must speak a rhotic dialect of English. Must pass a pure-tone hearing screening at 20dB hearing level. Must pass a brief examination of oral structure and function. Must exhibit less than 30% accuracy, based on consensus across 2 trained listeners, on a probe list eliciting rhotics in various phonetic contexts at the word level.

Must exhibit no more than 3 sounds other than /r/ in error on the Goldman-Fristoe Test of Articulation-3 (GFTA-3).

Exclusion Criteria:

Must not receive a T score more than 1.3 SD below the mean on the Wechsler Abbreviated Scale of Intelligence-2 (WASI-2) Matrix Reasoning Must not receive a scaled score of 7 or higher on the Recalling Sentences and Formulated Sentences subtests of the Clinical Evaluation of Language Fundamentals-5 (CELF-5).

Must not have an existing diagnosis of developmental disability or major neurobehavioral syndrome such as cerebral palsy, Down Syndrome, or Autism Spectrum Disorder

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in perceptually rated accuracy of /r/ | The timepoints for comparison will be from baseline to after both groups have completed 4 weeks of VAB and when both groups have completed the target 12 weeks of treatment (all types interventions: VAB, Perception training and no treatment).
  To assess generalization of treatment gains to untreated words, participants will be assessed with standard probes containing 45 syllables, 50 words and 5 sentences with rhotic targets in various phonetic contexts. Stimuli in each probe will be presented individually in randomized order with blocking by stimulus type (word, syllable, sentence). No auditory models will be provided; for children with reading difficulty, semantic cues will be provided to elicit the intended word.
  Individual words will be isolated from the audio record of each word probe and presented in randomized order for binary rating (correct/ incorrect) by 4 trained listeners who are blind to treatment condition and time point (but will see the written representation of each target word). We will use the proportion of "correct" ratings for each token as our primary measure of perceptually rated accuracy from which we will fit a multilevel model as the primary outcome variable.

SECONDARY OUTCOMES:
Socio-emotional well-being | Baseline and after all interventions are completed (target time frame: 12 weeks)
  This 11-item survey, which asks parents to report the impact of speech disorder on their child's social, emotional, and academic well-being, was validated in a published study by members of the research team [1]. An impact score, calculated as described in our previous research [1], will be used as the primary measure of socio-emotional well-being.
Percent accuracy pooled across Identification Perception task | The timepoints for comparison will be from baseline to after both groups have completed 4 weeks of VAB and when both groups have completed the target 12 weeks of treatment (all types interventions: VAB, Perception training and no treatment).
  Treatment task 2 (identification) is identical to the tasks used to assess performance in the baseline phase, with the single exception that accuracy feedback is provided during the treatment phase. In Task 2, accuracy in classifying stimuli as /r/ or / w/ will be assessed relative to the mean across responses from typical participants in our online participants from the previous funding cycle.
Percent accuracy pooled across Category Goodness Perception task | The timepoints for comparison will be from baseline to after both groups have completed 4 weeks of VAB and when both groups have completed the target 12 weeks of treatment (all types interventions: VAB, Perception training and no treatment).
  Treatment task 3 (category goodness judgment) are identical to the tasks used to assess performance in the baseline phase, with the single exception that accuracy feedback is provided during the treatment phase. In Task 3, accuracy in category goodness judgment will be assessed relative to the "gold-standard" ratings determined by consensus across at least four expert listeners.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Hitchcock, PhD, Principal Investigator — Montclair State University
Locations (1):
- Montclair State University, Montclair, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No